CLINICAL TRIAL: NCT04362787
Title: High Pressure Non Invasive Ventilation in Hypercapnic Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Eissa Helmy Abdelhafeez, Assistant Lecturer, Assiut University
Other Study IDs: High pressure
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Acute Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High pressure _ low pressure non-invasive ventilation: In the high-pressure NIV,52 patients will undergo pressure-limited NPPV at a higher IPAP level. IPAP is initially set at 20 cmH2O and continuously adjusted by increments and decrements of 1-2 cmH2O (up to 30 cmH2O), according to patients' tolerance, to obtain a tidal volume (VT) of 15 mL/kg of IBW.
  2- EPAP for patients with COPD will be started at EPAP 5 and will be increased till 7 and for the patients with hypoventilation syndrome will be increased up to EPAP 8.
  3-Respiratory rate 10-12 b/min.
  Interventions: Device: High pressure non invasive ventilation in acute hypercapnic respiratory failure

INTERVENTIONS:
Device: High pressure non invasive ventilation in acute hypercapnic respiratory failure — Usage of High pressure non invasive ventilation in acute hypercapnic respiratory failure

SUMMARY:
High pressure NIV is a pressure limited ventilation, stating IPAP pressure at 20 cmH2O and gradually increasing pressure up to 30 cmH2O according to patient tolerance.

DETAILED DESCRIPTION:
Noninvasive ventilation (NIV): refers to the administration of ventilatory support without using an invasive artificial airway (endotracheal tube or tracheostomy tube). NPPV is well established in the management of acute on chronic hypercapnic respiratory failure secondary to acute exacerbation of COPD (AECOPD), obesity hypoventilation syndrome, and restrictive thoracic disorders.

During the past years NIV was applied by using low pressure inspiratory positive airway pressure (IPAP), which means titrating inspiratory pressure starting at 10 cmH2O and increasing pressure gradually according to patient tolerance maximum up to 20 cm H2O.

There is still about 15% failure rate while using conventional low pressure NIV, this failure rate may be attributed to the following:

1. Still in a number of patients with conventional low pressure NIV, PaCO2, and pH worsen with subsequent deterioration and need for invasive ventilation.
2. Despite lowering PaCO2 value with conventional NIV ventilation but it is not normalized so with minimal derangement in clinical condition of the patient it worsens again.
3. Also abnormally high level PaCO2 may have a negative impact on vital organs.
4. Low pressure may be associated with patient intolerance , and discontinuation of NIV.

Recently high pressure NIV used aiming to improve outcome of NIV. High pressure NIV is a pressure limited ventilation, stating IPAP pressure at 20 cmH2O and gradually increasing pressure up to 30 cmH2O according to patient tolerance. High pressure NIV is expected to improve alveolar ventilation, decreasing dead space ventilation, and work of breathing, so it can improve the outcome result .

ELIGIBILITY:
Inclusion Criteria:

All patients admitted in Assiut University Hospital and Assiut Police Hospital with acute hypercapnic respiratory failure due to COPD and Obesity hypoventilation syndrome (OHS) indicated for conventional NIV.

Patients who failed on low pressure NIV will be shifted to high pressure NIV with any of these conditions:

1. PH <7.30 or less than admission level.
2. RR > 35b/m or more than admission level.
3. SpO2 < 88%.

Exclusion criteria: (4)

1. Age <18 years.
2. Excessive amount of respiratory secretions or weak cough.
3. Upper airway obstruction.
4. Recent oral, facial or cranial trauma or surgery.
5. Sever abdominal distension.
6. Active upper gastrointestinal bleeding.
7. Cardiac or respiratory arrest.
8. PH<7.25.
9. Arterial oxygen tension /fraction of inspired oxygen (PaO2 / FiO2) <150mmHg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who failed on low pressure NIV will be shifted to high pressure NIV with any of these
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
High pressure non invasive ventilation in acute hypercapnic respiratory failure | Patients will assessed after 2 hours from increasing pressure
  To study the efficacy of safety of high pressure NIV in acute hypercapnic respiratory failure due to COPD and obesity hypoventilation syndrome who refractory to low pressure NIV.
High pressure non invasive ventilation in acute hypercapnic respiratory failure | Patients will assessed after 2 hours from increasing pressure
  Effect of high pressure NIV on length of hospital stay , need for invasive mechanical ventilation, mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Hu Ahmed, Study Director — Professor of chest diseases Faculty of medicine Assiut university